CLINICAL TRIAL: NCT01610180
Title: Open Label Multicenter Study of Eltrombopag for the Treatment of Immune ThrombocytoPenia (ITP) Secondary to Chronic Lymphoproliferative Disorders (LPDs)
Brief Title: Eltrombopag for the Treatment of Immune ThrombocytoPenia (ITP) Secondary to Chronic Lymphoproliferative Disorders (LPDs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Progetto Ematologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VI-Plt-01
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic; Autoimmune Thrombocytopenic Purpura; Autoimmune Thrombocytopenia; Chronic Lymphocytic Leukemia; Non Hodgkin's Lymphoma
Keywords: Eltrombopag; ITP; LPD; leukemia; Immune ThrombocytoPenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Leukemia | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eltrombopag Olamine (Other): Eltrombopag Olamine Initial dose 50 mg/day for 14 days. Then adjusted according to platelet count
  Interventions: Drug: Eltrombopag Olamine

INTERVENTIONS:
Drug: Eltrombopag Olamine — Initial dose : 50 mg/day for 14 days.
  Next doses:
  1. If platelet count <60000/µL, increase daily dose by 25 mg to a maximum of 150 mg/day for next 14 days in 14 days courses. If response criteria not met after 14 days of the maximum dose stop treatment (no response).
  2. If platelet count >60000/µL and ≤200000/µL same dose for the next 14 days.
  3. If platelet count >200000/µL and ≤400000/µL decrease the daily dose by 25 mg. Wait 14 days to assess the effects of this and any subsequent dose adjustments.
  4. If platelet count >400000/µL, stop Eltrombopag; increase the frequency of platelet monitoring to twice weekly. Once the platelet count is <150000/µL, reinitiate therapy at a daily dose reduced by 25 mg.
  Other Names: Revolade; Eltrombopag

SUMMARY:
With conventional treatments (i.e. iv Ig, steroids) the overall response rate of ITP secondary to LPD is generally lower than in primary ITP, and usually not higher than 50% (95% CI 27-72). Eltrombopag which has proved very effective in primary ITP could be effective also in ITP secondary to LPDs.

This novel ITP specific treatment might spare these patients not only from bleeding risk but also from toxic or inappropriate cytotoxic therapies, not otherwise demanded by the burden of the underlying disease.

DETAILED DESCRIPTION:
The denomination of Chronic Lymphoproliferative Disorders (LPD) encompasses a variety of indolent lymphomas grouped into a single clinical category and, as such, this terminology is not included in the current WHO classification. With indolent lymphomas clinicians refer to those lymphomas not associated with an aggressive clinical course and in which often treatment can be delayed. Specifically the following lymphomas by the WHO classification will be considered among indolent lymphomas: small lymphocytic lymphoma/chronic lymphocytic leukemia, follicular lymphoma, marginal zone lymphoma, mantle cell lymphoma, lymphoplasmacytic lymphoma, hairy-cell leukemia, Hodgkin's lymphoma. In 1 to 5% of the different LPDs (lowest in follicular lymphoma, highest in chronic lymphocytic leukemia) a clinically relevant thrombocytopenia, often complicated by bleeding symptoms, may complicate the clinical course, frequently still when the tumor burden is low and not demanding treatment. This thrombocytopenia, when not accompanied by massive bone marrow tumor infiltration or not secondary to chemotherapeutic treatment, is thought to share an immune pathogenic mechanism similar to primary immune thrombocytopenia (ITP).

With conventional treatments (i.e. iv Ig, steroids) the overall response rate of ITP secondary to LPD is generally lower than in primary ITP, and usually not higher than 50% (95% CI 27-72). Therefore, any new treatment having a response rate above 50% but not inferior than 20% could be considered a promising treatment for ITP secondary to LPD. Furthermore, no significant platelet increase is expected without treatment in ITP secondary to LPD. Eltrombopag which has proved very effective in primary ITP could be effective also in ITP secondary to LPDs.

This novel ITP specific treatment might spare these patients not only from bleeding risk but also from toxic or inappropriate cytotoxic therapies, not otherwise demanded by the burden of the underlying disease.

Phase 2, single arm, open-label, prospective, multicenter, safety/efficacy study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of any of the following B-cell chronic LPD, as defined by WHO 2008 classification: small lymphocytic lymphoma/chronic lymphocytic leukemia, follicular lymphoma, marginal zone lymphoma, mantle cell lymphoma, lymphoplasmacytic lymphoma, hairy cell leukemia, Hodgkin's lymphoma.
2. Occurrence of ITP diagnosed on the basis of predefined criteria.
3. Not likely to necessitate any cytotoxic treatment for the following 6 months, according to clinical stage and performance status.
4. Platelet count less than 30,000/µL; patients with platelet count between 30 and 50,000/µL only in case of bleeding signs or symptoms.
5. Age greater than or equal to 18 years.
6. Absence of a personal or family (up to first degree relatives) history of venous or arterial thromboembolism.
7. ECOG performance status ≤2.
8. Adequate liver and renal function.
9. Absence of active Hepatitis B (HBsAg+ or HBV-DNA+), Hepatitis C (HCV-Ab+), or HIV infection.

9) Provided informed consent. 10) Negative pregnancy test or lactation 11) No antiplatelet or anticoagulant ongoing treatments

Exclusion Criteria:

1. Subjects with any clinically relevant abnormality, other than LPD or ITP, or any other medical condition or circumstance, which in the opinion of the investigator makes the subject unsuitable for participation in the study.
2. Subjects with any concurrent malignant disease other that the LPD and/or a recent history of cancer treatment with systemic chemotherapy and/or radiotherapy. Exception: Subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
3. Subjects with screening bone marrow fibers of either MF Grade 3 using European Consensus scale or Grade 4 using Bauermeister scale (see Appendix 1).
4. Subjects with a QTc >450 msec or > 480 msec for subjects with Bundle Branch Block.
5. Subjects with recent history of alcohol/drug abuse as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of responders to eltrombopag as defined by changes in the platelet count, in platelet transfusion requirements and/or in the bleeding symptoms during the 6 months of treatment. | 6 months of treatment for each patient
  Response criteria according to the International Working Group publication (Rodeghiero et al, Blood 2009).

SECONDARY OUTCOMES:
Assessment of the safety profile of eltrombopag in patients with LPD using the CTCAE criteria. | 9 months
  Adverse event reports graded with the National Cancer Institute Common Terminology Criteria for Adverse Events, version 3.0 and laboratory assessments at each on-treatment and post-treatment visit. Physical examination, general laboratory tests, including liver function tests, blood cell count and peripheral blood smear examination, flow cytometry at scheduled visits. Bone marrow biopsy, CT scan of the neck, chest and abdomen at enrollment, if not already done in the three preceding months, at the end of study and 3 months thereafter.
Number of patients meeting permanent discontinuation criteria | From enrollment to end of study duration (24 weeks) and of extension phase (up to 5 years after first patient enrollment)
  The following permanent discontinuation criteria were applied during the study and extension period: failure to respond; progression of the underlying disease demanding treatment; drug related toxicity or any adverse events ≥ grade 3 or peripheral blood and/or bone marrow findings suggesting marrow fibrosis (grade 3 or 4 of Bauermaister scale) or myelodisplasia or myeloproliferation including an increment of CD4 positive cell > 3 %.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Visco, MD, Principal Investigator — Department of Hematology, San Bortolo Hospital, Vicenza, Italy
Locations (1):
- Department of Hematology, Ospedale San Bortolo, Vicenza, Italy

REFERENCES:
- [Background] Visco C, Rodeghiero F. Immune thrombocytopenia in lymphoproliferative disorders. Hematol Oncol Clin North Am. 2009 Dec;23(6):1261-74. doi: 10.1016/j.hoc.2009.08.006. PMID 19932433
- [Background] Visco C, Ruggeri M, Laura Evangelista M, Stasi R, Zanotti R, Giaretta I, Ambrosetti A, Madeo D, Pizzolo G, Rodeghiero F. Impact of immune thrombocytopenia on the clinical course of chronic lymphocytic leukemia. Blood. 2008 Feb 1;111(3):1110-6. doi: 10.1182/blood-2007-09-111492. Epub 2007 Nov 6. PMID 17986663
- [Background] Visco C, Maura F, Tuana G, Agnelli L, Lionetti M, Fabris S, Novella E, Giaretta I, Reda G, Barcellini W, Baldini L, Neri A, Rodeghiero F, Cortelezzi A. Immune thrombocytopenia in patients with chronic lymphocytic leukemia is associated with stereotyped B-cell receptors. Clin Cancer Res. 2012 Apr 1;18(7):1870-8. doi: 10.1158/1078-0432.CCR-11-3019. Epub 2012 Feb 9. PMID 22322667
- [Derived] Visco C, Rodeghiero F, Romano A, Valeri F, Merli M, Quaresimini G, Volpetti S, Santi RM, Carli G, Lucchini E, Passamonti F, Rambaldi A, Motta G, Borchiellini A, d'Amore ESG, Ruggeri M. Eltrombopag for immune thrombocytopenia secondary to chronic lymphoproliferative disorders: a phase 2 multicenter study. Blood. 2019 Nov 14;134(20):1708-1711. doi: 10.1182/blood.2019001617. PMID 31570488